CLINICAL TRIAL: NCT00154219
Title: A 13-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Group Trial of Lumiracoxib (COX189) 100 mg o.d. in Patients With Primary Hip Osteoarthritis Using Celecoxib (200 mg o.d.) as a Positive Control
Brief Title: Efficacy and Safety Study of Lumiracoxib in Patients With Primary Hip Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2367
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis, Hip, Lumiracoxib, Efficacy, Safety
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — lumiracoxib; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Lumiracoxib (drug)

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability, and safety of the investigational drug, lumiracoxib as compared to celecoxib and placebo in subjects with hip osteoarthritis. Both lumiracoxib and celecoxib belong to the same class of drug (COX-2 selective nonsteroidal anti-inflammatory drugs [NSAIDs]).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary hip osteoarthritis
* Qualifying pain intensity in the hip joint
* Requiring NSAID therapy

Exclusion Criteria:

* Rheumatoid arthritis or other inflammatory joint disease
* Disease or disorder that may interfere with pain assessment of the hip
* Open knee/hip surgery within the last year
* Past history of heart attack, stroke or angina (chest pain)
* Liver disorder
* History of severe adverse reactions of any kind under lumiracoxib or celecoxib treatment

Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2004-11; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
WOMAC 3.1 LK questionnaire after 13 weeks of treatment
Patient's global assessment of disease activity (VAS) after 13 weeks of treatment

SECONDARY OUTCOMES:
Overall OA pain intensity (VAS)by visit
Physician's global assessment of disease activity (VAS) by visit
Response to treatment according to OARSI criteria by visit
Actual OA pain intensity at 12 hours post-dose by visit
Number of rescue tablets taken during the study

CONTACTS AND LOCATIONS:
Locations (5):
- For US Site Information, contact Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Various Sites, Multiple Cities, Canada
- Various Sites, Multiple Cities, Germany
- Various Sites, Multiple Cities, Italy
- Various Sites, Multiple Cities, United Kingdom

REFERENCES:
- [Derived] Schnitzer TJ, Dattani ID, Seriolo B, Schneider H, Moore A, Tseng L, Sallstig P, Rebuli R, Maxwell T. A 13-week, multicenter, randomized, double-blind study of lumiracoxib in hip osteoarthritis. Clin Rheumatol. 2011 Nov;30(11):1433-46. doi: 10.1007/s10067-011-1776-4. Epub 2011 May 24. PMID 21607551
- See also: Novartis patient recruitment website — http://www.osteoarthritistrial.com/